CLINICAL TRIAL: NCT05716139
Title: Preeclampsia Following Natural vs. Artificial Cycle Frozen Embryo Transfer
Brief Title: Natural Cycle vs Programmed Cycle Frozen Embryo Transfer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: As per institutional protocol unable to recruit adequate amount of participants
Sponsor: Indira IVF Hospital Pvt Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIHPL-UDR/RCT/013_2022
Record Dates: First submitted 2023-01-21; First posted 2023-02-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2023-07

CONDITIONS: Infertility; Frozen Embryo Transfer; Preeclampsia and Eclampsia
Keywords: Reproduction; In vitro fertilization; Natural Frozen Embryo Transfer; Artificial Frozen Embryo Transfer; Preeclampsia
MeSH Terms: conditions — Infertility; Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Intervention Model Description: Open labelled parallel group randomized Controlled Trial
Masking Description: Parallel group open labelled masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Natural Cycle (Active Comparator): In this,hCG trigger and Luteal Phase Support is monitored for the natural frozen embryo cycle procedure of IVF.
  Interventions: Procedure: Natural Cycle
- Artificial Cycle (Other): In this, endometrial preparation and Luteal Phase Support is monitored for the artificial frozen embryo cycle procedure of IVF.
  Interventions: Procedure: Artificial Cycle

INTERVENTIONS:
Procedure: Natural Cycle — The participant will be administered a S/C injection of 250mcg r-hCG to assist ovulation and timing of the embryo transfer, when the dominant follicle reaches ≥ 18mm and serum LH < 20 IU/L, the administration of r-hCG will be in the evening, and the embryo transfer will be scheduled seven days later (window of ± two days). The participant will begin transvaginal progesterone gel (8 %) twice daily starting 36 hrs after the trigger until ten weeks of gestation.
  Arms: Natural Cycle
Procedure: Artificial Cycle — Estrogen priming with oral estradiol valerate 6mg/day (2mg every 8 hours) starting from cycle D1-D5 after a first TVU. TVU will be performed 10-15 days after beginning estradiol until ET ≥ 7mm, maximum until 21 days. Patients will begin progesterone injection 100mg/day until blastocyst transfer. Frozen embryo transfer will be performed on day 6 +/- 2 days of progesterone administration. After embryo transfer, a supplementation with transvaginal progesterone gel (8 %) twice daily starting from the day of embryo transfer until ten weeks of gestation. Patients will continue Estradiol 2 mg thrice daily until 6 weeks of gestation; then dose tapering will be done to 2 mg twice daily until 9 wks of gestation. From 9th wk the estrogen dose will be tapered further to 2 mg once daily for 10 days before stopping.
  Arms: Artificial Cycle

SUMMARY:
The goal of this[ type of study: randomized controlled trial]is to compare Preeclampsia following Natural vs. Artificial Cycle in patients undergoing frozen embryo transfer.

The main question[s] it aims to answer is

• Does NC-FET decreases the incidence of preeclampsia in patients undergoing frozen embryo transfer as compared to AC-FET ?

The main objective is to compare the proportion of preeclampsia in women with a viable pregnancy with natural cycle protocol to artificial cycle protocol when practicing frozen embryo transfer. Participants recruited will be divided into two ARM(1513 per arm). ARM 1 will undergo the Natural Cycle procedure of Embryo transfer, and ARM 2 will undergo the Artificial Cycle procedure of Embryo transfer. The primary outcome will be the proportion of preeclampsia. The duration of the study is around 2 year.

DETAILED DESCRIPTION:
The Research question(PICO) addressed is Does NC-FET decreases the incidence of preeclampsia in patients undergoing frozen embryo transfer as compared to AC-FET . The hypothesis taken is NC-FET will decrease the incidence of preeclampsia compared to AC-FET. The sample size is taken as 3026 (1513 per arm). The Primary Objective is to compare the proportion of preeclampsia in women with a viable pregnancy with natural cycle protocol to artificial cycle protocol when practicing frozen embryo transfer. The study outcome of the proportion of preeclampsia after 20 weeks of gestation or 6 weeks post-delivery. There are two arms-Arm 1 Active Comparator: Natural Cycle and Arm 2 control: Artificial Cycle FET. The Randomization is done through Random Allocation as per computer generated sequence. The Blinding/masking is done Open labeled. The Study Duration is from Feb 2023 to Jan 2025. Participation Duration is 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial preparation with Hormone replacement therapy/ Natural cycle.
* Age 21-45 years following an autologous IVF cycle (with or without preimplantation genetic testing for aneuploidy)
* BMI > 18 and < 30 kg/m2
* Endometrial thickness ≥ 7 mm after estrogen therapy or on the day of ovulation
* Blastocyst embryo transfer

Exclusion Criteria:

* Uterine diseases (e.g. submucosal fibroids, polyps, previously diagnosed Müllerian abnormalities)
* Hydrosalpinx untreated.
* Recurrent pregnancy loss (≥ 3 previous miscarriages)
* Recurrent implantation failure (≥ 3 previously failed embryo transfers of good-quality blastocysts)
* Allergy to study medication
* Pregnancy or lactation at recruitment
* Contraindications for hormonal treatment

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 172 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
proportion of preeclampsia | after the 20th week of gestation up to six weeks postpartum
  The primary efficacy endpoint is the proportion of preeclampsia in women assigned to a natural cycle protocol compared to the proportion of preeclampsia in women assigned to an artificial cycle protocol.

SECONDARY OUTCOMES:
Biochemical Pregnancy Rate | 6 weeks after Embryo Transfer
  Pregnancies diagnosed only by β-human chorionic gonadotropin detection without a gestational sac visualized by vaginal ultrasound at the 6th gestational week.
Implantation Rate | 4 weeks +2 weeks after ET
  The number of gestational sacs observed by transvaginal ultrasound at the 6th gestational week per the number of embryos transferred.
Clinical Pregnancy Rate | 4 weeks +2 weeks after ET
  Detection of a foetal heartbeat on transvaginal ultrasound at the 6th gestational week per embryo transfer cycle.
Ongoing Pregnancy Rate | 12 weeks after embryo Transfer
  Presence of gestational sacs with a heartbeat at the 12th gestational week per embryo transfer cycle.
Live Birth Rate | 28 weeks(+12 weeks) after embryo transfer
  The number of deliveries that resulted in at least one live birth per 100 Embryo transferred cycle.
Miscarriage Rate | Within 20 weeks of gestation
  Number of spontaneous pregnancy losses in which a gestational sac/s was previously observed (before 20th gestational weeks) per 100 clinical pregnancy.
Preterm birth | < 37 weeks
  Preterm is defined as babies born alive before 37 weeks of pregnancy are completed
Extreme preterm birth | 20-28 weeks
  Extreme Preterm is defined as babies born alive before 28 weeks of pregnancy
Fetal growth restriction | 20-40 weeks of gestation
  Fetal growth restriction (FGR) is most often defined as an estimated fetal weight less than the 10th percentile for gestational age by prenatal ultrasound evaluation
Fetal birthweight | within 30 minutes of birth
  Is defined as the weight of baby just after birth
Premature detachment of normally inserted placenta | 12 weeks of GA till labor
  It is defined as a premature separation of the placenta before delivery.
Maternal hypertension | After 20 weeks of GA till 6 weeks postpartum
  It is defined as blood pressure more than 140/90 mm Hg detected first time after 20 weeks of gestation till 6 weeks of postpartum without proteinuria
Eclampsia | After 20 weeks of GA till 6 weeks postpartum
  Eclampsia is defined as the new onset of generalized tonic-clonic seizures in a woman with preeclampsia.
HELLP Syndrome | After 20 weeks of GA till 6 weeks postpartum
  It is defined as hemodialysis, elevated liver enzymes, and low platelet count
Maternal mortality | from start of pregnancy to 42 weeks of pregnancy
  Maternal death is defined as pregnancy or its management (excluding accidental or incidental causes) during pregnancy and childbirth or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy
Fetal death | 20 weeks of GA before delivery
  Fetal death refers to the spontaneous intrauterine death of a fetus after 20 weeks of GA before delivery
Frequency of adverse events | through study completion, an average of 1 year
  An adverse event (AE) is any untoward medical occurrence in a patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Indira IVF Hospital Private Limited, Udaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers after publication of primary results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After six months of publication of primary results statistical plan and ICF
Access Criteria: IPD will be shared on request

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists' Committee on Obstetric Practice; Committee on Genetics; U.S. Food and Drug Administration. Committee Opinion No 671: Perinatal Risks Associated With Assisted Reproductive Technology. Obstet Gynecol. 2016 Sep;128(3):e61-8. doi: 10.1097/AOG.0000000000001643. PMID 27548556
- [Background] Baksh S, Casper A, Christianson MS, Devine K, Doody KJ, Ehrhardt S, Hansen KR, Lathi RB, Timbo F, Usadi R, Vitek W, Shade DM, Segars J, Baker VL; NatPro Study Group. Natural vs. programmed cycles for frozen embryo transfer: study protocol for an investigator-initiated, randomized, controlled, multicenter clinical trial. Trials. 2021 Sep 27;22(1):660. doi: 10.1186/s13063-021-05637-3. PMID 34579768
- [Background] Busnelli A, Schirripa I, Fedele F, Bulfoni A, Levi-Setti PE. Obstetric and perinatal outcomes following programmed compared to natural frozen-thawed embryo transfer cycles: a systematic review and meta-analysis. Hum Reprod. 2022 Jun 30;37(7):1619-1641. doi: 10.1093/humrep/deac073. PMID 35553678
- [Background] Devroey P, Polyzos NP, Blockeel C. An OHSS-Free Clinic by segmentation of IVF treatment. Hum Reprod. 2011 Oct;26(10):2593-7. doi: 10.1093/humrep/der251. Epub 2011 Aug 9. PMID 21828116
- [Background] Ginstrom Ernstad E, Wennerholm UB, Khatibi A, Petzold M, Bergh C. Neonatal and maternal outcome after frozen embryo transfer: Increased risks in programmed cycles. Am J Obstet Gynecol. 2019 Aug;221(2):126.e1-126.e18. doi: 10.1016/j.ajog.2019.03.010. Epub 2019 Mar 22. PMID 30910545
- [Background] Kawwass JF, Badell ML. Maternal and Fetal Risk Associated With Assisted Reproductive Technology. Obstet Gynecol. 2018 Sep;132(3):763-772. doi: 10.1097/AOG.0000000000002786. PMID 30095760
- [Background] Lee JC, Badell ML, Kawwass JF. The impact of endometrial preparation for frozen embryo transfer on maternal and neonatal outcomes: a review. Reprod Biol Endocrinol. 2022 Feb 28;20(1):40. doi: 10.1186/s12958-021-00869-z. PMID 35227270
- [Background] Luke B. Pregnancy and birth outcomes in couples with infertility with and without assisted reproductive technology: with an emphasis on US population-based studies. Am J Obstet Gynecol. 2017 Sep;217(3):270-281. doi: 10.1016/j.ajog.2017.03.012. Epub 2017 Mar 18. PMID 28322775
- [Background] Malik A, Jee B, Gupta SK. Preeclampsia: Disease biology and burden, its management strategies with reference to India. Pregnancy Hypertens. 2019 Jan;15:23-31. doi: 10.1016/j.preghy.2018.10.011. Epub 2018 Nov 2. PMID 30825923
- [Background] Rienzi L, Gracia C, Maggiulli R, LaBarbera AR, Kaser DJ, Ubaldi FM, Vanderpoel S, Racowsky C. Oocyte, embryo and blastocyst cryopreservation in ART: systematic review and meta-analysis comparing slow-freezing versus vitrification to produce evidence for the development of global guidance. Hum Reprod Update. 2017 Mar 1;23(2):139-155. doi: 10.1093/humupd/dmw038. PMID 27827818
- [Background] von Versen-Hoynck F, Schaub AM, Chi YY, Chiu KH, Liu J, Lingis M, Stan Williams R, Rhoton-Vlasak A, Nichols WW, Fleischmann RR, Zhang W, Winn VD, Segal MS, Conrad KP, Baker VL. Increased Preeclampsia Risk and Reduced Aortic Compliance With In Vitro Fertilization Cycles in the Absence of a Corpus Luteum. Hypertension. 2019 Mar;73(3):640-649. doi: 10.1161/HYPERTENSIONAHA.118.12043. PMID 30636552
- [Background] Chen JZ, Sheehan PM, Brennecke SP, Keogh RJ. Vessel remodelling, pregnancy hormones and extravillous trophoblast function. Mol Cell Endocrinol. 2012 Feb 26;349(2):138-44. doi: 10.1016/j.mce.2011.10.014. Epub 2011 Oct 25. PMID 22051447
- [Background] Shi Y, Sun Y, Hao C, Zhang H, Wei D, Zhang Y, Zhu Y, Deng X, Qi X, Li H, Ma X, Ren H, Wang Y, Zhang D, Wang B, Liu F, Wu Q, Wang Z, Bai H, Li Y, Zhou Y, Sun M, Liu H, Li J, Zhang L, Chen X, Zhang S, Sun X, Legro RS, Chen ZJ. Transfer of Fresh versus Frozen Embryos in Ovulatory Women. N Engl J Med. 2018 Jan 11;378(2):126-136. doi: 10.1056/NEJMoa1705334. PMID 29320646